CLINICAL TRIAL: NCT03570905
Title: Radiographic and Clinical Comparison of Post-reduction Splinting Constructs in the Treatment of Acute Displaced Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01697
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Radius Fractures
Keywords: acute, displaced distal radius fracture
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugartong Splint (Experimental)
  Interventions: Other: Sugar Tong Splint
- Clam Shell Splint (Experimental)
  Interventions: Other: Clam Shell Splint

INTERVENTIONS:
Other: Sugar Tong Splint — A splint made of 8-10 layers of plaster rolled into a single long sheet which begins at the distal volar crease of the hand and traverses around the elbow and stops at the dorsal metacarpal heads. The skin is protected with cotton cast padding (webril) and the splint is held in place with ace bandages
  Arms: Sugartong Splint
Other: Clam Shell Splint — A 2-part splint made of 8-10 layers of plaster. The piece traverses from the distal volar crease of the hand to the volar aspect of the proximal forearm. The second piece runs along the dorsal aspect of forearm from metacarpal heads to proximal forearm. The elbow is left free. In the same fashion as the sugar tong splint, the skin is protected with cotton cast padding (webril) and held in place with ace wrap
  Arms: Clam Shell Splint

SUMMARY:
Subjects with acute, displaced distal radius fractures will be randomized at the time of emergency room evaluation to one of two commonly accepted splinting methods for displaced distal radius fractures: sugar tong splints or volar/dorsal clam shell splints. Reduction will be performed in the usual, standard fashion and the selected splint applied. Standard radiographic measurements of alignment, including radial height, volar tilt and inclination will be measured on pre- and post- reduction radiographs by a single reviewer- who will be blinded to splint application type. At the first fracture follow-up visit, typically occurring between 5-10 days, as in standard practice, repeat radiographs of the wrist will be taken, and the same reviewer will measure alignment. As a secondary outcome, patients will also complete the disabilities of the arm, shoulder and hand (DASH) questionnaire at this visit, to compare patients' ability to perform activities of daily living with their respective splints.

ELIGIBILITY:
Inclusion Criteria:

* acute, displaced distal radius fracture
* isolated injury

Exclusion Criteria:

* polytrauma
* non-displaced fracture
* prior wrist fracture

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Displacement of fracture, measured by radial height | 1 Week
  >2 mm of radial height lost from immediate post-reduction radiographs
  A t-test will be performed with a p value < 0.05 to determine significance in loss of reduction A t-test will also be performed comparing individual parameters between the 2 splinting methods
Displacement of fracture, measured by volar tilt | 1 Week
  > 5 degrees of radial inclination lost from immediate post-reduction radiographs
  A t-test will be performed with a p value < 0.05 to determine significance in loss of reduction A t-test will also be performed comparing individual parameters between the 2 splinting methods
Displacement of fracture, measured by radial inclination | 1 Week
  > 10 degrees of volar tilt lost from immediate post-reduction radiographs
  A t-test will be performed with a p value < 0.05 to determine significance in loss of reduction A t-test will also be performed comparing individual parameters between the 2 splinting methods
Disabilities of the Arm, Shoulder,and Hand (DASH) outcome score | 1 Week
  30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nirmal Tejwani, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication. Researchers who provide a methodologically sound proposal will have access.
Access Criteria: Requests should be directed to nicole.stevens@nyumc.org. To gain access, data requestors will need to sign a data access agreement.